CLINICAL TRIAL: NCT00594178
Title: Palliative Strategies in Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Edgar Garcia-Rill, Director, Center for Translational Neuroscience
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24179; PRN # 12903 NIH
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2010-12

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Exercise group
  Interventions: Device: Motorized bicycle exercise training

INTERVENTIONS:
Device: Motorized bicycle exercise training — Passive exercise with a bicycle to bilateral legs. 5 days per week for 3 months

SUMMARY:
Spinal cord injury (SCI) leads to muscle atrophy, hyperreflexia and spasticity, symptoms that decrease quality of life and prevent effective rehabilitation. Previous findings from our labs found that a passive cycling exercise program, motorized bicycle exercise training (MBET), in adult spinally transected animals reduced muscle atrophy and normalized hyperreflexia. We found that MBET could prevent the onset of hyperreflexia after spinal transaction, that MBET could also be used to rescue from hyperreflexia once it had set in, and that MBET could induce savings in normalization of reflexes after MBET ceased. We also demonstrated that MBET was effective in rescuing from hyperreflexia in a chronic ASIA B SCI patient, and that short-term MBET could lead to brief savings in normalization of reflexes once MBET ceased. The proposed studies will test the ability to MBET to prevent the onset of hyperreflexia in a group of acute SCI patients trained before hyperreflexia has had a chance to set in. In addition, the proposed research will attempt to confirm the possibility that long-term MBET in chronic SCI patients will rescue from hyperreflexia once it has set in, and also produce significant savings in normalization of reflexes if carried out for long periods of time. We will also test the possibility that MBET in acute and/or chronic SCI patients could reduce or prevent muscle atrophy. The experimental design calls for assessing muscle mass using MRI scans, bone density using Dual-Energy X-ray Absortiometry (DEXA) scans, spasticity measures and electrophysiological measurements to determine low frequency habituation of the H-reflex. Assessments will be carried out before MBET, during a 25 week MBET block of time, and during a 12 week post MBET monitoring period. Changes in muscle mass, bone density, spasticity scales and H-reflex habituation will be compared across these interventions and between treated SCI victims and a group of control acute and chronic SCI victims undergoing standard of care during the same period.

ELIGIBILITY:
Inclusion Criteria:

* 1. An incomplete spinal cord injury at a level of C4 to T12.
* 2. 18 to 70 years of age.

Exclusion Criteria:

* 1. Joint contractures and/or spasticity that would hamper upright posture or use of MBET
* 2. A documented blood clot in the lower extremities
* 3. A history of lower extremity fractures (excludes randomization to the PWBT).
* 4. Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-10; Primary Completion 2008-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S. Kiser, MD, Principal Investigator — Center for Translational Neuroscience, UAMS; Edgar Garcia-Rill, PhD, Study Director — Center for Translational Neuroscience, UAMS
Locations (1):
- Center for Translational Neuroscience #847, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from my outpatient and inpatient clinical service who had a spinal cord injury starting on 4/1/2003 and ending on 3/9/2010
Pre-assignment Details: Patients were excluded from the study if we were unable to obtain an H-reflex on nerve conduction study due to this being the primary endpoint we were assessing.
Groups:
- Passive Exercise With Motorized Bicycle: The exercise was conducted from the subjects wheelchair with the feet attached to the bicycle by velcro straps and extra ankle dorsiflexion, provided by wedges on the pedal, to stretch the gastrocnemeus and soleus muscles. 60 minutes of exercise at with a goal of 60 rpm per training session. The exercise was conducted three times a week for 16 weeks or 5 times a week for 12 weeks, for an average of 50 sessions. Each subjects bone density and lean muscle mass was measured by DEXA scan, using a low radiation dose to determine the effect of exercise by comparing the subjects change in both parameters before the exercise and then after the exercise.
Period: Overall Study
Arm/Group | Passive Exercise With Motorized Bicycle
Started | 17
Completed | 12
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Passive Exercise With Motorized Bicycle
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.38 (14.4314)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Muscle Mass Via Dual-Energy X-ray Absortiometry (DEXA)Scan Data
Description: Lean muscle mass was measured with Dual-Energy X-ray Absortiometry (DEXA) scan, which uses low dose radiation to assess bone density and soft tissue density. pre and post, three month exercise protocol on a passivie motorized exercise bicycle.
Time Frame: baseline and 3 months
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Passive Exercise With Motorized Bicycle
Number analyzed (Participants) | 12
grams
  Baseline | 6104.45 (1087.6)
  Post exercise | 6355.3 (1667.8)
Statistical Analysis 1: Comparison: Passive Exercise With Motorized Bicycle; Paired samples T-test was used to assess the statisical changes between baseline and post-exercise lean muscle mass; Test type: Superiority or Other; p = .318, t-test, 2 sided; Mean Difference (Final Values) = -250.8, 95% CI 2-sided [-778.87 to 277.21]

2. Secondary Outcome: Bone Density Via Dual-Energy X-ray Absortiometry (DEXA) Scan
Description: Bone mineral density was measured with Dual-Energy X-ray Absortiometry (DEXA) scan pre and post, three month exercise protocol on a passive motorized exercise bicycle.
Time Frame: baseline and 3 months Post-exercise
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Passive Exercise With Motorized Bicycle
Number analyzed (Participants) | 12
grams/cm^2
  Baseline | 1.134 (.29041)
  3 months post exercise | 1.069 (.25988)
Statistical Analysis 1: Comparison: Passive Exercise With Motorized Bicycle; Paired samples T-test was used to assess the statisical changes between baseline and post-exercise bone density; Test type: Superiority or Other; p = .011, t-test, 2 sided; Mean Difference (Final Values) = .0645, 95% CI 2-sided [.01827 to .11073]

ADVERSE EVENTS:
Arm/Group | Passive Exercise With Motorized Bicycle
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
This was a pilot study to determine if a passive exercise bicycle would suppress the H-reflex after a spinal cord injury. We were not able to collect stable H-reflex data. However, the Dual-Energy X-ray Absortiometry (DEXA) scan data was useable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No